CLINICAL TRIAL: NCT03908801
Title: Evaluation of Specialized Water Dance Intervention (SWAN) for Individuals With Profound Intellectual and Multiple Disabilities: A Randomized Controlled Trial.
Brief Title: Evaluation of Specialized Water Dance Intervention
Acronym: SWAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Region Gävleborg (Other); Värmland County Council, Sweden (Other Government); Region Östergötland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18RS788/RÖL
Record Dates: First submitted 2019-03-19; First posted 2019-04-09 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2020-10

CONDITIONS: Spastic; Pain, Chronic; Stress; Quality of Life
MeSH Terms: conditions — Muscle Spasticity; Chronic Pain

STUDY DESIGN:
Intervention Model Description: The participants are first randomized to the intervention or control group and when the intervention for the first group is completed, the intervention is given to the second group (former control group). Since the prevalence of profound intellectual and multiple disabilities is low, the project is carried out as a multicenter study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Specialized water dance intervention
  Interventions: Behavioral: Specialized water dance intervention
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Specialized water dance intervention — Group activity in a warm pool (32-34 °C) led by two SWAN leaders. During each session, nine songs are played and the participants, assisted by a support person, perform dance movements rhythmically to the mood of the music. The songs are chosen to stimulate different movement patterns and to emphasize different emotions.
  Arms: Intervention

SUMMARY:
Individuals with profound intellectual and multiple disabilities (PIMD) have extensive health problems and need for personal assistance throughout the day. Few physical- and health promoting activities are available for them and among the activities, few have been scientifically evaluated. Specialized water dance intervention (SWAN) is a new method developed to relieve discomfort and promote physical wellbeing among people with PIMD. The aim of the study is to evaluate the effects of SWAN on stress, spasticity, pain, alertness, wellbeing and social interaction among individuals with PIMD.

Individuals with profound intellectual and multiple disabilities (PIMD) have extensive health problems and need for personal assistance throughout the day. Few physical and health promoting activities are available for them. Among the activities, few have been scientifically evaluated. Specialized water dance intervention (SWAN) is a new method developed to relieve discomfort and promote physical wellbeing among people with PIMD. The aim of the study is to evaluate the effects of SWAN on stress, spasticity, pain, alertness, wellbeing and social interaction among individuals with PIMD.

Prospective randomized controlled intervention study in which the effects of SWAN are tested in a two-group cross-over design with pre-, under- and post-measurements. The study is conducted as a multicenter study with four participating county councils/regions I Sweden (Varmland County Council, Region Orebro County, Region Ostergotland and Region Gavleborg).

The SWAN intervention is given once a week for 3 months (12 occasions). Each SWAN session is 45 minutes and is led by two SWAN leaders.

ELIGIBILITY:
Inclusion Criteria:

* have a profound intellectual and multiple disabilities corresponding to level IV-V in the Gross Motor Function Classification System.
* aged 16-65 years
* be accustomed to water and not find discomfort of activities in water.

Exclusion Criteria:

* severe hearing impairment/deafness
* have wounds/infections that are infectious in the pool

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Stress | 14 weeks
  Cortisol in saliva
Spasticity | 14 weeks
  The Modified Ashworth Scale is used to assess muscle tone. The flexor muscles of the elbows and the extensor muscles of the knees on the participants left and right side are tested. The muscle tone is scored on a 6-point scale from 0 (No increase in muscle tone) to 5 (Affected part(s) is(are) rigid in flexion or extension). The higher the score, the more resistance to passive movement.
Wellbeing: Observed (questionnaire) | 12 weeks
  The questionnaire includes items on spasticity, anxiety, pain, social interaction and joy. The support person assess the patients' level of spasticity, anxiety, pain, social interaction and joy three times: before, during and after each session. Each item is assessed on a five-point Likert scale, from 'not at all present' (1) to 'present all the time' (5). The research group has developed the questionnaire.
Quality of Life assessment: EQ5D | 14 weeks
  Quality of life was assessed using the proxy version of the EuroQol Five Dimension (EQ5D). The EQ5D is divided into five items: mobility, self-care, Daily activities, pain and discomfort, anxiety and depression. The items are scored on a 5 point scale, as well as a visual analogue scale ranging from 0 (worst imaginable health) to 100 (best imaginable health).

SECONDARY OUTCOMES:
Behavior | 12 weeks
  Video assisted observation. Each person will be video recorded in the pool on three occasions (1st, 6th and 12th session). The responsible intervention leader and the project coordinator perform the video recording. From the video recordings, assessments are made of the patient's expression of emotions and social interaction, through a structured assessment protocol developed by the research group. The video material is transferred to the computer and encoded according to a pre-established protocol using a computer program-coding tool.
Goal attainment | 14 weeks
  We use the Goal Attainment Scaling (GAS), which provides an individualized, criterion-referenced measure of change. The GAS procedure involves: (a) defining a unique set of goals for each participant, (b) specifying a range of possible outcomes for each goal (on a scale recommended to contain five levels, from -2 (the participants baseline level before the intervention) to +2(represent much better than expected after the intervention) and (c) using the scale to evaluate the participants change after a specified intervention period.
Muscular pain | 12 weeks
  Observed (video).Each person will be video recorded in the pool on three occasions (1st, 6th and 12th session). The video recording is performed by the responsible intervention leader and the project coordinator. From the video recordings, assessments are made of the patient's expression of pain, through a structured assessment protocol developed by the research group. The video material is transferred to the computer and encoded according to a pre-established protocol using a computer program-coding tool.

OTHER OUTCOMES:
Experience of implementation of study intervention | 2 years
  Interviews with assistants, intervention leaders and head of organisations.

CONTACTS AND LOCATIONS:
Overall Officials: Mats G Karlsson, Professor, Study Chair — Region Örebro County
Locations (1):
- University Health Care Research Center, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lundqvist LO, Materne M, Frank A, Morelius E, Duberg A. Salivary cortisol levels and stress in adults with profound intellectual and multiple disabilities participating in the Structured Water Dance Intervention: a randomised controlled crossover trial. Sci Rep. 2022 Oct 19;12(1):17418. doi: 10.1038/s41598-022-21573-x. PMID 36261594
- [Derived] Granberg A, Materne M, Lundqvist LO, Duberg A. Navigating change - managers' experience of implementation processes in disability health care: a qualitative study. BMC Health Serv Res. 2021 Jun 10;21(1):571. doi: 10.1186/s12913-021-06570-6. PMID 34112151
- See also: Description of the SWAN project — https://www.researchweb.org/is/fourol/project/240151